CLINICAL TRIAL: NCT03558360
Title: Preoperative Dry Lean Body Mass as a Prognostic Factor for Excess Weight Loss After Bariatric Surgery.
Acronym: MMS-CB
Status: Unknown | Type: Observational
Last Known Status: Recruiting
Sponsor: Centre Hospitalier Departemental Vendee (Other)
Responsible Party: Sponsor
Other Study IDs: CHD 048-17
Record Dates: First submitted 2018-06-04; First posted 2018-06-15 (Actual); Last update posted 2021-12-23 (Actual); Status verified 2021-12

CONDITIONS: Bariatric Surgery Candidate
Keywords: lean body mass; bariatric surgery

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Cross-Sectional
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (1):
- Bariatric surger: Bariatric surgery and impedance measurement
  Interventions: Diagnostic Test: Impedance measurement

INTERVENTIONS:
Diagnostic Test: Impedance measurement — Measurement of dry lean body mass berfore bariatric surgery by impedance measurement.

SUMMARY:
Bariatric surgery is currently the only method that has proven long-term effectiveness in obesity. Although the benefit of physical activity on weight loss has been demonstrated, no correlation has ever been reported between preoperative lean body mass and postoperative weight loss. Dry lean mass is probably an essential prognostic factor for the effectiveness of bariatric surgery.

The main objective of this study is to define a preoperative dry lean body mass threshold as a worst prognostic factor for weight loss one year after bariatric surgery.

The management of patients included in this study was modelled on the management usually offered to patients followed for the same pathology in the diabeto-endocrinology department. There are no study-specific examinations that are not part of current practice.

ELIGIBILITY:
Inclusion Criteria:

* BMI ≥ 40 or BMI ≥ 35 kg/m2 and a complication that can be improved after bariatric surgery: cardiovascular disease including hypertension, severe metabolic disorder including type 2 diabetes, sleep apnea syndrome or other severe respiratory disorder, hepatic steatosis, disabling osteoarticular disease.
* Patient requiring bariatric surgery (sleeve-gastrectomy or gastric bypass)
* Patient who has agreed to participate in the study
* Patient with social security coverage.

Exclusion Criteria:

* Patient with a contraindication to bariatric surgery (cognitive or psychological disorders, severe eating disorders, addiction to alcohol or psychoactive substances, contraindication to general anaesthesia, multiple history of digestive surgery, high risk of undernutrition (progressive cancer, chronic inflammatory bowel disease, cirrhosis, severe renal insufficiency...)
* Pregnant or lactating women
* Minor patient
* Major patient under tutorship, curatorship, or deprived of liberty
* Patient unable to understand protocol and / or give express consent
* Patient not affiliated with a social security system or beneficiary of such a scheme
* Patient participating in an intervention-type clinical research protocol likely to modify the evaluations of this protocol
* adults under the protection of justice

Ages: 18 Years to 65 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: Patients presenting (or having presented since 2014) an obesity with a bariatric surgery project and followed by endocrinologist doctors.
Sampling Method: Non-Probability Sample
Enrollment: 180 (Estimated)
Dates: Start 2018-10-15 (Actual); Primary Completion 2022-04-01 (Estimated); Study Completion 2022-09-01 (Estimated)

PRIMARY OUTCOMES:
Measurement of dry lean mass in pre-operative by impedance measurement | 12 months after bariatric surgery
  Excess weight loss at M12: ideal weight is defined in relation to height for a BMI of 25.0 kg/m2. Excess weight is the difference between the observed weight and the ideal weight. Excess weight loss is the ratio of weight loss to excess weight.

CONTACTS AND LOCATIONS:
Overall Officials: Barbara FEIGEL-GUILLER, MD, Study Director — Centre Hospitalier Départemental Vendée
Locations (1):
- Centre Hospitalier Departemental Vendée, La Roche-sur-Yon, France